CLINICAL TRIAL: NCT07381205
Title: Prospective Evaluation of Transplant Associated Thrombotic Microangiopathy (TA-TMA) Markers in a High-risk Cohort of Adults Undergoing Allogeneic Stem Cell Transplantation (SCT)
Brief Title: Assessing the Incidence of Transplant Associated Thrombotic Microangiopathy (TA-TMA) in Adult Patients Undergoing Allogeneic Stem Cell Transplant (SCT)
Status: Not yet recruiting | Type: Observational
Sponsor: Manuel Ricardo Espinoza-Gutarra (Other)
Collaborators: BMS Foundation (Unknown); Viracor Eurofins (Unknown)
Responsible Party: Sponsor-Investigator, Manuel Ricardo Espinoza-Gutarra, Assistant Professor, University of Alabama at Birmingham
Organization: University of Alabama at Birmingham (Other)
Other Study IDs: UAB2537
Record Dates: First submitted 2026-01-08; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Transplant Associated Microangiopathy TAM; Transplant Complication
Keywords: Transplant Associated Thrombotic Microangiopathy; Allogeneic Stem Cell Transplant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral Blood Bone Marrow Aspirate
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort 1: Main Cohort of patients who fulfill Inclusion Criteria
- Cohort 2: Patients who develop GVHD with any of the following characteristics and were not included in cohort 1
  1. Grade III-IV aGVHD, or SR-aGVHD of any grade, whichever occurs first
  2. Moderate to Severe cGVHD or SR-cGVHD of any grade, whichever occurs first
- Cohort 3: Patients included in either cohort 1 or 2 who are diagnosed with TA-TMA and receive eculizumab

SUMMARY:
The goal of this observational study is to learn about the incidence of Transplant Associated Thrombotich Microangiopathy (TA-TMA), which is a known but underreported complication of Allogeneic Stem Cell Transplant (SCT). The main question it aims to answer is:

What is the incidence of TA-TMA in adults undergoing SCT? How does TA-TMA diagnosis impact survival and other outcomes? Patients undergoing SCT will be eligible for this study, which will consist of collection of biological samples and standard clinical follow up.

DETAILED DESCRIPTION:
This will be a prospective non-interventional study that will include patients undergoing allogeneic stem cell transplant (SCT) deemed to be at high risk for developing Transplant Associated Thrombotic Microangiopathy (TA-TMA). All patients will have prospective biospecimens collected per study schedule starting prior to SCT. Biospecimens will be collected for use in translational testing and sent to Viracor for commercial testing. Results of commercial testing will be made available to treating physicians. Diagnosis of TA-TMA will be made based on clinical and laboratory values according to existing consensus guidelines, however, therapeutic decisions will be left up to the treating clinical team. Patients will be followed up for clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  1. Adult male or female, age ≥18
  2. Undergoing allogeneic SCT at UAB for any indication and any donor source.
  3. For patients in cohort 1: Patients deemed high-risk for developing high-risk TA-TMA as stated by any of the following criteria*:

     1. BMI > 35[42]
     2. Mismatched donor (either Haploidentical or Mismatched Unrelated donor)[18, 29]
     3. Non-Malignant Transplant Indication (Severe Aplastic Anemia or Sickle Cell Disease)[18, 43]
     4. Acute Lymphoblastic Leukemia (any kind)[18, 31]
     5. African American, Hispanic, Asian or Native American Ethnicity [44]
     6. Myeloablative Conditioning Regimen[18]
     7. Pre-Existing Renal Disease** (defined as any of the following: 24 Hr Creatinine Clearance <60, baseline serum creatinine > 1.2, 24 hr proteinuria >150mg or random spot urine Protein Creatinine ratio > 150mg/g)[20, 45]
     8. TBI-containing conditioning regimen >400cGy [46]
     9. Prior Autologous or Allogeneic SCT[45]

        * *Some of these criteria have been adapted from pediatric literature due to a higher number of publications in that setting and in cases where the adult data is lacking or contradictory.
        * **Proteinuria thresholds are obtained from KDIGO guidelines and include moderate and severe levels of proteinuria[47].
  4. Females of childbearing potential must have a negative urine or serum pregnancy test prior to enrollment.
  5. For patients in cohort 2: Patients who develop GVHD with any of the following characteristics and were not included in cohort 1

     1. Grade III-IV aGVHD, or SR-aGVHD of any grade, whichever occurs first
     2. Moderate to Severe cGVHD or SR-cGVHD of any grade, whichever occurs first
  6. For patients in cohort 3: Patients included in either cohort 1 or 2 who are diagnosed with TA-TMA and receive eculizumab

Exclusion Criteria:

* Exclusion Criteria

  1. Any other active malignancy requiring treatment or with expected survival ≤1 year.
  2. Patients with psychiatric illness or social situations that would limit compliance with the study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing allogeneic stem cell transplant (SCT) deemed to be at high risk for developing Transplant Associated Thrombotic Microangiopathy (TA-TMA) as per inclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 85 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Primary Objectives | From enrollment until 1 year post SCT
  The primary objective of the study is to report the rates of high-risk TA-TMA in a cohort for high-risk patients undergoing allogeneic SCT. High-risk TA-TMA will be defined as per the ASTCT Harmonization Criteria which will include the TMA Harmonization panel consensus recommended diagnostic criteria and any of the high-risk TA-TMA features (Schoettler et al. TCT March 2023).
Co-Primary Objective | From enrollment until 1 year post SCT
  To evaluate rates of Non-Relapse Mortality (NRM) in patients with and without TA-TMA. NRM is defined as the rate of death from any cause in patients who do not exhibit any sign of relapse or progression of their underlying hematologic malignancy

SECONDARY OUTCOMES:
Secondary Objectives | From enrollment until 1 year post SCT
  * To evaluate rates of Overall Survival (OS) in patients with and without high-risk TA-TMA
  * OS is defined as the time from the date of SCT until death.
Secondary Objective | From enrollment until 1 year post SCT
  -To evaluate rates of Graft Versus Host Free Relapse Free Survival (GFRS) in patients with and without high-risk TA-TMA.
  GRFS is defined as the time from the date of SCT until occurrence of grade III-IV aGVHD, and or cGVHD requiring systemic immune suppression, and or disease progression or death whichever comes first.
Secondary Objective | From enrollment until 1 year post SCT
  -To validate previously described risk factors and prognostic scores for the development of high-risk TA-TMA -We will compare other prognostic markers that have been described in the literature such as EASIX score, degree of proteinuria among others to evaluate their correlation with rate and severity of TA-TMA
Secondary Objective | From enrollment until 1 year post SCT
  -To evaluate kinetics of sC5b-9 in patients with and without high-risk TA-TMA -These analytes will be obtained as per study procedure and their changes will be described.

OTHER OUTCOMES:
Exploratory Objectives | From enrollment until 1 year post SCT
  -To evaluate the impact of therapeutic interventions by treating physicians on biomarkers and clinical outcomes These analytes will be obtained as per study procedure and their changes will be described both in isolation and in association with prespecified variables
Exploratory Objective | From enrollment until 1 year post SCT
  -To evaluate the association between high-risk TA-TMA development and relapse. Relapse is defined as the rate of patients having their underlying hematologic malignancy relapse or progress after SCT
Exploratory Objective | From enrollment until 1 year post SCT
  To evaluate, using cohort 3, the association between CH50 levels, eculizumab through levels and high-risk TA-TMA response to eculizumab treatment. These analytes will be obtained as per study procedure and their changes will be described both in isolation and in association with other, pre-specified, variables
Exploratory Objective | From enrollment until 1 year post SCT
  -To evaluate Patient Reported Outcomes (PROs) in patients with and without high-risk TA-TMA PROs will be obtained at pre-determined times for all patients in the study, the results will be reported descriptively.

CONTACTS AND LOCATIONS:
Locations (1):
- O'Neal Comprehensive Cancer Center at UAB, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No